CLINICAL TRIAL: NCT05316051
Title: Effect of Different Foot Orthosis Inverted Angles on Walking Kinematics in Females With Flexible Flatfeet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nour Mustafaalsaafin (Other)
Responsible Party: Sponsor-Investigator, Nour Mustafaalsaafin, Postgraduate Student, University of Sharjah
Organization: University of Sharjah (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: u20105881
Record Dates: First submitted 2022-03-19; First posted 2022-04-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Flexible Flatfoot
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 25° inverted angle foot orthoses (Experimental)
  Interventions: Device: Inverted foot orthoses
- 15° inverted angle foot orthoses (Experimental)
  Interventions: Device: Inverted foot orthoses
- Control (No Intervention)

INTERVENTIONS:
Device: Inverted foot orthoses — Inverted functional orthoses will be used in this study based on Blake (1986) inverted orthotic technique. Two groups of foot orthosis will be fabricated with two different inverted angles: 25° inverted angle and 15° inverted angle.
  Arms: 15° inverted angle foot orthoses; 25° inverted angle foot orthoses

SUMMARY:
Inverted orthosis is a type of rigid foot orthosis that was designed to aid in controlling high degrees of foot pronation. It is essential to administer patients foot orthoses with different inverted angles, with higher angles prescribed when greater reduction of foot pronation is indicated. However, there is shortage of clinical knowledge regarding the inverted angle in terms of biomechanical changes. The aim of this study is to investigate the effect of different inverted angles of foot orthoses on the walking kinematics in females with flexible flatfeet.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Within the age group of 18-35 years
* Asymptomatic flexible flatfeet
* Resting Calcaneal Stance Position angle of ≥ 4° in valgus in both feet (bilateral)

Exclusion Criteria:

* Previous surgery of the lower limbs or spine that might affect the performance of the study procedures
* Any severe medical or musculoskeletal conditions that may have affected the lower limbs
* Fixed flatfoot deformity
* Leg length discrepancy (> 1cm)
* Pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Lower limb kinematics | Through study completion, an average of 1 year.
  Lower limb kinematics will be processed and calculated using a motion capture system (SMART-DX, BTS Bioengineering, Milan, Italy). The following kinematic variables will be obtained for each subject : (i) maximum hip extension angle, (ii) maximum hip adduction angle, (iii) maximum hip external rotation angle, (iv) maximum knee flexion angle during loading response, (v) maximum knee extension angle during midstance, (vi) maximum knee flexion angle at toe off, (vii) minimum knee abduction angle, (viii) maximum knee abduction angle, (ix) maximum knee external rotation angle, (x) maximum knee internal rotation angle, (xi) maximum ankle plantarflexion angle during loading response, (xii) maximum ankle dorsiflexion angle during midstance, (xiii) maximum ankle plantarflexion angle at toe off, (xiv) maximum ankle external rotation angle, (xv) maximum ankle internal rotation angle.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma A. Hegazy, PhD, Principal Investigator — University of Sharjah
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No